CLINICAL TRIAL: NCT02271828
Title: Clinically Node Negative Breast Cancer Patients Undergoing Breast Conserving Therapy: Sentinel Lymph Node Procedure Versus Follow-Up.
Brief Title: Omitting Sentinel Node Procedure in Breast Cancer Patients Undergoing Breast Conserving Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Borstkanker Onderzoek Groep (Network); Dutch Cancer Society (Other); Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOOG 2013-08; BOOG 2013-08 (Other: Dutch Breast Cancer Trialists' Group (BOOG)); KWF UM 2014-6679 (Other Grant/Funding Number: The Dutch Cancer Society (KWF))
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sentinel lymph node procedure (Active Comparator): Sentinel lymph node procedure according to the Dutch breast cancer guideline
  Interventions: Procedure: Sentinel lymph node procedure
- No sentinel lymph node procedure (No Intervention): No sentinel lymph node procedure

INTERVENTIONS:
Procedure: Sentinel lymph node procedure — Sentinel lymph node procedure according to the Dutch breast cancer guideline
  Arms: Sentinel lymph node procedure

SUMMARY:
STUDY AIM To decrease the number of breast cancer patients receiving over treatment of the axilla, in order to positively influence the axillary morbidity rate and quality of life.

PRIMARY OBJECTIVE To determine whether omitting the sentinel lymph node procedure is not inferior to the current axillary staging regimen in clinically node negative breast cancer patients undergoing breast conserving therapy, in terms of regional recurrence rate.

HYPOTHESIS The sentinel lymph node procedure can be safely omitted in clinically node negative breast cancer patients undergoing breast conserving therapy. This will lead to a decreased axillary morbidity rate, with a non-inferior regional recurrence-, distant-disease free- and overall survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 years or older
* Pathologically confirmed invasive breast carcinoma
* A clinical T1-2 tumor
* Will be treated with lumpectomy and whole breast radiotherapy
* Clinically node negative status: no signs of axillary lymph node metastases at physical examination and preoperative axillary ultrasound (or negative cyto-/histopathology)
* Written informed consent

Exclusion Criteria:

* Clinically node positive pre-operative
* Bilateral breast cancer
* Evidence of metastatic disease
* History of invasive breast cancer
* Previous treatment of the axilla with surgery or radiotherapy (except surgery for hidradenitis suppurativa or for other superficially located skin lesions, such as naevi)
* Pregnant or nursing
* Other prior malignancies within the past 5 years (except successfully treated basal cell and squamous cell skin cancer, carcinoma in situ of the cervix or carcinoma in situ of the ipsilateral or contralateral breast) or unsuccessfully treated malignancies > 5 years before randomization
* Unable or unwilling to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1644 (Estimated)
Dates: Start 2015-04; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Regional recurrence rate | Up to ten years
  Regional recurrence is defined as tumour recurrence and as residual tumour that became clinically apparent in ipsilateral axillary, infraclavicular and supraclavicular lymph nodes (pathologically proven).

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein L Smidt, MD, PhD, Principal Investigator — Maastricht University Medical Centre, Maastricht, the Netherlands; Hans JW de Wilt, MD, PhD, Principal Investigator — Radboud University Medical Centre, Nijmegen, the Netherlands
Locations (22):
- Netherlands (22):
  - Maastricht University Medical Centre+, Maastricht, Limburg
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - Flevoziekenhuis, Almere Stad
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Rijnstate, Arnhem
  - Amphia ziekenhuis, Breda
  - Deventer ziekenhuis, Deventer
  - Catharina ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Groene Hart ziekenhuis, Gouda
  - UMC Groningen, Groningen
  - Spaarne Gasthuis, Haarlem
  - Alrijne, Leiden
  - St. Antonius ziekenhuis, Nieuwegein
  - Canisius-Wilhelmina ziekenhuis, Nijmegen
  - Radboud UMC, Nijmegen
  - Laurentius ziekenhuis, Roermond
  - Haga ziekenhuis, The Hague
  - Diakonessenhuis, Utrecht
  - UMC Utrecht, Utrecht
  - Zuwehofpoort ziekenhuis, Woerden
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Wintraecken VM, van Roozendaal LM, Simons JM, de Vries J, van Kuijk SMJ, Vane MLG, van Dalen T, Sackey H, van der Hage JA, Strobbe LJA, Linn SC, Lobbes MBI, Poortmans PMP, Tjan-Heijnen VCG, van de Vijver KKBT, Westenberg HH, Dirksen CD, de Wilt JHW, Boersma LJ, Smidt ML. Three-year patient-reported outcomes of the BOOG 2013-08 RCT evaluating omission of sentinel lymph node biopsy in early-stage breast cancer patients treated with breast conserving surgery: Impact of personality traits on health-related quality of life. Br J Surg. 2025 Apr 30;112(5):znaf031. doi: 10.1093/bjs/znaf031. PMID 40365927
- [Derived] van Roozendaal LM, Vane MLG, van Dalen T, van der Hage JA, Strobbe LJA, Boersma LJ, Linn SC, Lobbes MBI, Poortmans PMP, Tjan-Heijnen VCG, Van de Vijver KKBT, de Vries J, Westenberg AH, Kessels AGH, de Wilt JHW, Smidt ML. Clinically node negative breast cancer patients undergoing breast conserving therapy, sentinel lymph node procedure versus follow-up: a Dutch randomized controlled multicentre trial (BOOG 2013-08). BMC Cancer. 2017 Jul 1;17(1):459. doi: 10.1186/s12885-017-3443-x. PMID 28668073
- See also: Study description BOOG study center — https://www.boogstudycenter.nl/studie/273/2013-08-lumpectomie.html